CLINICAL TRIAL: NCT05133934
Title: Investigation of Traditional Chinese and Western Medicine in the Real World of Knee Osteoarthritis: A Multicenter Cohort Study
Brief Title: Traditional Chinese and Western Medicine for Knee Osteoarthritis
Acronym: TCMWMKOA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Guanghua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine (Unknown); Yueyang Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai University of TCM (Unknown); China-Japan Friendship Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); Henan Provincial People's Hospital (Other); Jiangsu Province Hospital of Traditional Chinese Medicine (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Affiliated Hospital of Nanjing University of Chinese Medicine (Other); Traditional Chinese Medicine Hospital of Xinjiang Uygur Autonomous Region (Unknown); First Affiliated Hospital of Heilongjiang Chinese Medicine University (Other); Integrated Hospital of Traditional Chinese Medicine, Southern Medical University (Unknown); Ruijin Hospital (Other); The Second Clinical Medical College of Zhejiang University of Traditional Chinese Medicine (Unknown); Affiliated Hospital of Shandong University of Traditional Chinese Medicine (Other); Southwest Hospital, China (Other); The Second People's Hospital Affiliated to Fujian University of Traditional Chinese Medicine (Unknown); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); ShuGuang Hospital (Other); Shanghai Municipal Hospital of Traditional Chinese Medicine Affiliated to Shanghai University of TCM (Unknown); Shanghai University of Traditional Chinese Medicine (Other); Dongzhimen Hospital, Beijing (Other); Nanfang Hospital, Southern Medical University (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Zhong Lidan, Assistant Professor, Hong Kong Baptist University
Other Study IDs: TCMWM-KOA
Record Dates: First submitted 2021-08-12; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — A cohort study will be used to collect patient data, analyze the clinical characteristics, TCM syndromes, and treatment of knee osteoarthritis in China

SUMMARY:
A cohort study will be used to collect patient data, analyze the clinical characteristics, traditional Chinese medicine (TCM) syndromes, and treatment of knee osteoarthritis (KOA) in China to accumulate clinical data and clarify the status of KOA in the real world background. It will lay a clinical foundation for further study of KOA in the future, and bring certain clinical value for Chinese patients with KOA.

DETAILED DESCRIPTION:
This is a multicenter cohort study. It is planned to carry out multicenter investigation and research on the current situation of knee osteoarthritis in the real world, conduct large-scale investigation on the clinical population of patients with knee osteoarthritis, and establish a research, quality control, data management and statistical analysis platform for the clinical practical application of knee osteoarthritis and hospital registration. This study aims to discover the current clinical characteristics, TCM syndromes, and treatment status of patients with knee osteoarthritis in China, and provide reliable data support for the clinical treatment of KOA. It is estimated that 5000 patients from 23 centers across China will be recruited. Various demographic and disease-related information will be documented, including name, gender, age, job category, disease course, medical consultation experience, treatment satisfaction and so on. Patients will also complete a series of scales, containing Visual Analog Scale (VAS) Score, Knee Injury and Osteoarthritis Outcome Score (KOOS), Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index, 9-item patient health questionnaire (PHQ-9), SF-12 quality of life, TCM syndrome score sheet, etc. The primary outcome will be the pain (rest pain) VAS, KOOS, WOMAC knee osteoarthritis index score and TCM syndrome score. Secondary outcomes include patient's knee joint function examination, X-ray examination results, blood routine, biochemical indicators and pharmacoeconomic data.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has repeated knee joint pain in the past month;
2. X-ray film (standing position or weight-bearing position) shows narrowing of the joint space, subchondral bone sclerosis and/or cystic degeneration, and osteophyte formation on the joint edges;
3. Age ≥50 years old;
4. Morning stiffness time ≤30min;
5. There is bone friction sound (sensation) during activity.

Patients who meet the diagnostic criteria 1 + (any 2 of 2, 3, 4, 5) can be diagnosed as KOA.

Exclusion Criteria:

Patients who do not meet the diagnostic criteria for knee osteoarthritis

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 5000 patients who meet the diagnostic criteria for knee osteoarthritis from the 23 affiliated hospitals/centers across China will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Patient-assessed Pain (rest pain) Visual Analog Scale (VAS) score | 1 month
  The pain VAS is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, 10 centimeters (100 mm) in length, each end of this scale is an extreme label of the symptom, "no pain" (corresponding to the scale of 0) and "pain too intense to be tolerated" (corresponding to the scale of 100). Respondents indicate their degree of acceptance to a statement by specifying a point on the continuous scale in between two endpoints.
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100.
  A higher score indicates greater pain intensity.
The Knee Injury and Osteoarthritis Outcome Score (KOOS) | 1 month
  KOOS is a self-administered, knee-specific instrument to assess the patients' opinion about their knee and associated problems.
  The KOOS evaluates both short-term and long-term consequences of knee injury. It holds 42 items in 5 separately scored subscales:
  * Symptoms & Stiffness (7 items)
  * Pain (9 items)
  * Function in daily living (ADL Function) (17 items)
  * Sport and Recreation Function (5 items)
  * Quality of Life (4 items)
  A Likert scale is used and all items have 5 possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the 5 scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopedic assessment scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
WOMAC Knee Osteoarthritis Index Score | 1 month
  WOMAC knee osteoarthritis index is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  * Pain (5 items):
  * Stiffness (2 items):
  * Physical Function (17 items)
  A Likert scale is used and all items have 5 possible answer options: none (0), mild (1), moderate (2), severe (3), and extreme (4).
  A total WOMAC score is created by summing the items for all three subscales (0-96), and higher scores indicate worse pain, stiffness, and functional limitations.
TCM Syndrome Differentiation and Symptom Score | 1 month
  Patients' health as characterized by CM diagnostic pattern & clinical characteristics is recorded using the standard of TCM syndrome differentiation that adopts the 2019 Chinese Society of Chinese Medicine Clinical Diagnosis and Treatment Guidelines for TCM Orthopedics and Traumatology - Knee Arthritis (Knee Osteoarthritis) Syndrome Differentiation Standard (cold-damp arthralgia syndrome, damp-heat arthralgia syndrome, stagnation of Qi and blood stasis syndrome, liver and kidney deficiency syndrome, and qi and blood weakness syndrome)

SECONDARY OUTCOMES:
Knee Joint Function | 1 month
  knee joint's function Questionnaire
Morning Stiffness Time (in minutes) | 1 month
  Morning stiffness time (in minutes) is self recorded by patients daily when they wake up in the morning, to assess the severity of the stiffness.
  Prolonged morning stiffness that lasts more than an hour and up to several hours suggest worsened osteoarthritis or other inflammatory types of arthritis.
9-Item Patient Health Questionnaire (PHQ-9), | 1 month
  PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression.
  The severity of depression is categorized into mild, moderate, moderately severe and severe depression. The final question on the PHQ-9 screens for the presence and duration of suicide ideation.
12-Item Short Form Survey (SF-12) for Quality of Life of Patients | 1 month
  The SF-12 is a self-reported quality of life measure to be scored by a researcher, to assess the impact of health on patients' everyday life, and keeps track of how patients feel and how well they are able to do their usual activities.
  It consists of 12 questions measuring eight domains of health, including physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. These health domain scores are aggregated into the physical component summary (PCS) score and the mental component summary (MCS) score.
  Higher component summary scores indicate better health and better health-related quality of life (HRQoL).
Complete blood count (CBC) | 1 month
  CBC is done to help evaluate red and white blood cells and hemoglobin, and to monitor the side effects of some OA treatments
C-reactive Protein (CRP) | 1 month
  CRP is done to detect inflammation and test for the activity of the disease; an increased level of CRP suggests other forms of inflammatory arthritis, such as rheumatoid arthritis (RA) instead of osteoarthritis.
Erythrocyte Sedimentation Rate (ESR) | 1 month
  The ESR rate increases as a result of any cause or focus of inflammation. ESR is done to detect inflammation in the body; ESR will be increased in other forms of inflammatory arthritis, such as RA but not in osteoarthritis.
Liver Function | 1 month
  Liver function test is done to assess patients' liver function, as abnormal liver function tests are often seen in patients with inflammatory arthritis.
Kidney Function | 1 month
  Kidney function test is done to assess patients' kidney function, as kidney toxicity is a potential side effect of some arthritis medications.
Urine Routine | 1 month
  Urine test is done to assess patients' kidney function, as kidney toxicity is a potential side effect of some arthritis medications.
Examination of X-Ray | 1 month
  X-rays of the affected knee joints to assess the loss of cartilage, bone damage, bone spurs, and narrowing of the joint space using following grading scale:
  * Grade 0 (normal)
  * Grade I (suspicious narrowing of joint space, possibly osteophytes)
  * Grade II (obvious osteophytes, slightly narrowed joint space)
  * Grade III (moderate osteophytes, more obviously narrowed joint space, slightly sclerotic subchondral bone)
  * Grade IV (large number of osteophytes, significantly narrowed joint space, extremely obvious sclerosis changes, joints hypertrophy and obvious deformities)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Zhong, MD, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- Hong Kong, Kowloon Tong, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided